CLINICAL TRIAL: NCT04432480
Title: Parasympathetic Activity Evaluation by Newborn Infant Parasympathetic Evaluation (NIPE) Monitor (MDMSTM, Loos, France) During Routine General Anesthesia in Children
Brief Title: NIPE Monitoring Values During Routine Pediatric Anesthesia
Acronym: OMNIPED
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_31; 2020-A00059-30 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia; Nociceptive Pain
Keywords: General anesthesia; Nociceptive Pain; Monitoring; Pediatric anesthesia
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children: 0-15 years old children undergoing surgery under general anesthesia
  Interventions: Procedure: NIPE (Newborn Infant Parasympathetic Evaluation) monitoring

INTERVENTIONS:
Procedure: NIPE (Newborn Infant Parasympathetic Evaluation) monitoring — Non invasive monitor connected to standard anesthesia monitor (no part of the device in contact with the patient) during anesthesia.

SUMMARY:
Description of the standard values and fluctuations of the new NIPE index during routine pediatric anesthesia. NIPE monitor connected to anesthesia monitor, displays an instantaneous value ranging from 0 to 100. NIPE values described at different time points during anesthesia: beginning of induction, intubation, extubation, skin incision, opioid administration, vasopressors or atropine administration, transfusion, volume expansion. In addition, NIPE values during hemodynamic events (heart rate or blood pressure increase greater than 20%) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Surgery under general anesthesia
* Absence of analgesic treatment in the 24 hours before the intervention

Exclusion Criteria:

* Central or peripheral neuropathy
* Non sinus arrythmia, pace maker
* Cardiac surgery
* Analgesic medication within 24 hours before surgery
* Anti cholinergic or anti arrythmic chronic medication
* Opposition of the legal tutor or of the child

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children in the pediatric surgical wardof:
  * Lille University hospital (Lille, France)
  * Armand Trousseau Hospital (Paris, France)
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Variation of the instantaneous NIPE index after opioid administration | 5 minutes after opioid administration

SECONDARY OUTCOMES:
the area under the ROC curve of NIPE value | Baseline and 5 minutes before the first hemodynamic event.
  the NIPE value is definied by the predictibility of a hemodynamic event : 20% increase in Baseline heart rate, blood pressure and NIPE values recorded just before skin incision
Variation of the instantaneous NIPE index after skin incision | 5 minutes after skin incision
Variation of the instantaneous NIPE index after insertion of airway control device | 5 minutes after insertion of airway control device
Variation of the instantaneous NIPE index after removal of airway control device | 5 minutes after removal of airway control device
Variation of the instantaneous NIPE index after anesthetic induction | 5 minutes after anesthetic induction

CONTACTS AND LOCATIONS:
Overall Officials: Anne LAFFARGUE, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France